CLINICAL TRIAL: NCT05903092
Title: A Phase II Trial of MOnaliZumab in Combination With durvAlumab (MEDI4736) Plus Platinum-based chemotheRapy for First-line Treatment of Extensive Stage Small Cell Lung Cancer (MOZART)
Brief Title: MOnaliZumab in Combination With durvAlumab (MEDI4736) Plus Platinum-based chemotheRapy for First-line Treatment of Extensive Stage Small Cell Lung Cancer
Acronym: MOZART
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Cohort A fully accrued; pending addition of a Cohort B.
Sponsor: Hirva Mamdani (Other)
Collaborators: AstraZeneca (Industry); Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Hirva Mamdani, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN21-530
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer; SCLC; Extensive Stage Small Cell Lung Cancer
Keywords: Small cell lung cancer; First-line therapy; Chemoimmunotherapy; Immunotherapy; Monalizumab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; monalizumab; Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Durvalumab + Monalizumab + Chemotherapy (Experimental): On Day 1 of every Cycle for the first 4 Cycles (Cycle = 21 Days):
  Durvalumab 1500mg IV, Monalizumab 1500mg IV, Either Carboplatin AUC 5-6 OR Cisplatin 75-80mg/m^2
  On Days 1-3 of every Cycle for the first 4 Cycles:
  Etoposide 80-100mg/m^2
  On Day 1 of Cycles 5+ (Cycle = 28 Days):
  Durvalumab 1500mg IV Monalizumab 1500mg IV
  Interventions: Drug: Durvalumab; Drug: Monalizumab; Drug: Carboplatin or Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Durvalumab — 1500mg IV on Day 1 of every Cycle
  Other Names: Imfinzi
Drug: Monalizumab — 1500mg IV on Day 1 of every Cycle
Drug: Carboplatin or Cisplatin — On Day 1 of Cycles 1-4 by IV:
  Carboplatin: AUC 5-6 OR Cisplatin: 75-80mg/m^2
Drug: Etoposide — 80-100mg/m^2 IV on Days 1-3 of Cycles 1-4
  Other Names: VP-16

SUMMARY:
The study treatment will consist of a platinum drug (carboplatin or cisplatin per investigator's choice) plus etoposide plus durvalumab plus monalizumab every 3 weeks for 4 cycles. After 4 cycles, subjects will continue maintenance treatment with durvalumab plus monalizumab every 4 weeks until disease progression, unacceptable toxicity, decision to stop study treatment, or withdrawal of consent. Patients who have received one prior cycle of treatment before enrolling on the study will receive a total of 4 cycles with monalizumab, durvalumab, and chemotherapy. There will be a safety lead-in phase, including 6 to 12 patients, to confirm the safety of the proposed dose of monalizumab to use in combination with chemotherapy and durvalumab.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. Note: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0-2.
4. Histologically or cytologically confirmed diagnosis of small cell lung cancer:

   * Extensive disease (American Joint Committee on Cancer Stage (8th edition) IV SCLC [T any, N any, M1 a/b]), or
   * T3-4 disease due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan.
5. No prior systemic therapy for small-cell lung cancer, with the following exceptions:

   --Up to one cycle of platinum doublet chemotherapy with or without durvalumab is allowed up to 4 weeks prior to registration on this study. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab and monalizumab may be included only after consultation with the sponsor-investigator. Patients should not have received trilaciclib.
6. Measurable disease according to RECIST v1.1
7. Subjects with treated brain metastasis and those with untreated asymptomatic brain metastasis are eligible if they are clinically stable per investigator discretion and not requiring systemic steroids for ≥ 7 days. Prophylactic cranial radiation (PCI) is allowed per investigator's discretion.
8. Demonstrate adequate organ function. All screening labs to be obtained within 28 days prior to registration.

   * Absolute Neutrophil Count (ANC) > 1500mm^3
   * Hemoglobin ≥ 9 g/dL
   * Platelet Count (PLT) ≥ 100,000 per mm3
   * Calculated creatinine clearance ≥ 40 mL/min
   * Bilirubin ≤ 1.5 × upper limit of normal (ULN); subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), may be allowed with sponsor-investigator approval.
   * Apsartate aminotransferase (AST) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
   * Alanine aminotransferase (ALT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
9. Females of childbearing potential must have a negative serum pregnancy test at screening.
10. Females of childbearing potential and male subjects must be willing to abstain from heterosexual intercourse or to use an effective method(s) of contraception.
11. Life expectancy of ≥ 12 weeks.
12. Patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable through PCR to be eligible for this trial. Testing is not required for screening unless mandated by local authorities. Local guidelines for testing should be followed.

Exclusion Criteria:

1. Body weight ≤ 40 kg.
2. Receipt of radiotherapy to the chest within 6 months prior to initiating systemic therapy or planned consolidation chest radiation therapy. NOTE: Radiation therapy outside of the chest for palliative care (e.g., bone metastasis) is allowed but must be completed before the first dose of the study medication.
3. Active infection requiring intravenous antibiotic therapy.
4. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
5. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of study treatment. NOTE: Local surgery of isolated lesions for palliative intent is acceptable.
6. History of active primary immunodeficiency.
7. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
8. Presence of neurologic paraneoplastic syndrome.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., ulcerative colitis or Crohn's disease], systemic lupus erythematosus, sarcoidosis, Wegener syndrome [granulomatosis with polyangiitis], rheumatoid arthritis, hypophysitis, uveitis, etc). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 2 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
10. Current or prior use of immunosuppressive medication within 7 days before the first dose of monalizumab and 'on-study' durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication), and for prevention of chemotherapy induced nausea/vomiting per institutional standards.
11. Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment. NOTE: Subjects, if enrolled, should not receive live vaccine whilst receiving study treatment and up to 30 days after the last dose of study treatment.
12. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
13. Patients who have received prior one dose of durvalumab along with chemotherapy:

    * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    * Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤ Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
14. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
15. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per investigator discretion.
16. History of leptomeningeal carcinomatosis.
17. History of allogeneic organ transplantation.
18. Treatment with any investigational drug within 28 days prior to registration or concurrent enrolment in another clinical study, unless observational in nature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2028-01-03 (Estimated)

PRIMARY OUTCOMES:
1 year Progression Free Survival (PFS) | 1 year
  PFS is defined as the time from Day 1 of treatment (i.e., Day 1 of the first cycle of systemic therapy for SCLC, on study or initiated prior to enrolling on the study, whichever occurs first) until the criteria for disease progression is met as defined by RECIST 1.1 or death as a result of any cause.
Safety and Tolerability | 24 Months
  Safety and tolerability will be assessed by the grading of adverse events based on Common Toxicity Criteria for Adverse Events (CTCAE) v5.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 Months
  The objective response rate is the proportion of all subjects with confirmed PR or CR according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment)
Overall Survival (OS) | 24 Months
  OS is defined as the time from Day 1 of treatment (i.e., Day 1 of the first cycle of systemic therapy for SCLC, on study or initiated prior to enrolling on the study, whichever occurs first) until death as a result of any cause.
Intracranial PFS (iPFS) | 24 Months
  iPFS is defined as the time from Day 1 of treatment (i.e., Day 1 of the first cycle of systemic therapy for SCLC, on study or initiated prior to enrolling on the study, whichever occurs first) until the criteria for intracranial disease progression is met as defined by RECIST 1.1 or administration of brain radiation or death as a result of any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Hirva Mamdani, MD, Principal Investigator — Wayne State University
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Karmanos Cancer Center (Wayne State University), Detroit, Michigan
  - University of Virginia Health System, Charlottesville, Virginia